CLINICAL TRIAL: NCT00428168
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Examine the Effect of Betahistine on Body Weight Gain Due to Olanzapine Treatment
Brief Title: Study to Examine the Effect of Betahistine on Body Weight Gain Due to Olanzapine Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim Analysis result indicated the study will not show a significant benefit of the study medication on the primary endpoint.
Sponsor: OBEcure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BET202
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Weight Gain
Keywords: Betahistine; Weight Gain Control; Weight Gain due to Olanzapine Treatment; Obesity; Schizophrenic disorder
MeSH Terms: conditions — Weight Gain; Obesity; Schizophrenia | interventions — Betahistine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betahistine 24 mg (Experimental)
  Interventions: Drug: Betahistine
- Placebo (Placebo Comparator)
  Interventions: Drug: Betahistine

INTERVENTIONS:
Drug: Betahistine — Betahistine 24mg BID

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, multinational study. Approximately 78 subjects (39 per treatment group) will be randomized into this 16 week study.

A screening visit will be used to determine subject suitability for inclusion in the trial.

Within 7 days of the screening visit, subjects who meet all inclusion criteria and none of the exclusion criteria will be randomly assigned to 1 of the following 2 treatment groups:

* Olanzapine OD plus betahistine 24 mg BID (48 mg/day total),
* Olanzapine OD plus matching placebo BID.

Double-blind treatment will continue for 16 weeks. During this period, olanzapine dosage will be determined according to the discretion of the treating physician. In addition, 5 study visits (at 2, 4, 8, 12, and 16 weeks) will take place. Study medication (betahistine or matching placebo) will be administered BID (in the morning and together with olanzapine in the evening).

The primary statistical hypothesis to be tested is that the mean change from Baseline to Week 16 will be different between the treatment and placebo groups

ELIGIBILITY:
Inclusion Criteria:

* Subject (or legal guardian) is capable and willing to provide signed written informed consent;
* Male or female subjects 16 to 45 years of age;
* Body mass index in the range of 18.5 to 35 kg/m2;
* Diagnosed as having schizophrenia, schizoaffective disorder, schizophreniform disorder or a psychosis disorder that is not otherwise specified (NOS) according to the DSM-IV criteria;
* Maximum of 6 weeks cumulative lifetime exposure to risperidone, OR maximum of 3 weeks cumulative lifetime exposure to any other antipsychotic medication;
* Designated by the managing physician to be appropriate for treatment with olanzapine; and
* If female: is non-lactating, has a negative blood serum pregnancy test result, and does not plan on becoming pregnant during the study, or is not of childbearing potential (hysterectomy or tubal ligation at least 6 months prior to randomization or post-menopausal for 1 year); if of childbearing potential (including peri-menopausal women who have had a menstrual period within one year), must practice and be willing to continue to practice appropriate birth control (such as implants, injectables, oral contraceptives, intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire study duration.

Exclusion Criteria:

* Has obesity of known endocrine origin (e.g., Cushing's disease, Addison's disease, hypothalamic tumor);
* Has a medical history (e.g., morbid childhood obesity) and/or physical characteristics (e.g., polydactyly) suggestive of genetic obesity (e.g., ob/ob genotype) or syndromatic obesity (e.g., Prader-Willi syndrome, Bardet Biedl syndrome);
* Previous surgical procedures for weight loss;
* Has had liposuction within 1 year before screening or is planning to have liposuction during the study;
* Has a clinically significant history or presence of any of the following conditions:
* Active or past history of cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities;
* Type 1 diabetes mellitus;
* Type 2 diabetes mellitus with treatment other than metformin monotherapy and/or diet with HbA1c >8%;
* Severe type 2 diabetes with history of ketoacidosis or diabetic ulcers, or presence of retinopathy, neuropathy, or nephropathy;
* Renal insufficiency defined as a serum creatinine >=1.5 mg/dL (133 µmol/L) at screening;
* Malignant disease, other than basal cell carcinoma, within 5 years of screening;
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 x ULN;
* Thyroid-stimulating hormone (TSH) outside of the normal range;
* Plans on having any surgery (elective or otherwise) during the course of the study;
* Has uncontrolled hypertension (sitting blood pressure >160/95 mmHg at screening or randomization), uncontrolled hyperlipidemia (triglycerides [TG] >=400 mg/dL or low-density lipoprotein cholesterol [LDL] >160 mg/dL), or uncontrolled diabetes (HbA1c >8%);
* Diagnosis of asthma;
* History of peptic ulcers;
* History of HIV;
* Has a physical examination or electrocardiogram (ECG) with significant abnormalities, as judged by the investigator;
* Chronic antihistamine use or use of antihistamines within 14 days of randomization;
* History of pheochromocytoma
* Requires treatment with any of the following medications but has not been on a stable treatment regimen for a minimum of 90 days prior to screening:
* Hormone replacement therapy;
* Oral contraceptives;
* Antihypertensive agents;
* Metformin;
* Lipid-lowering agents; or
* Thyroid replacement therapy;
* Has been treated over the past 60 days, is currently treated, or is expected to require or undergo treatment with any of the following excluded medications;
* All prescription or over-the-counter agents taken for the purpose of weight reduction, including (but not limited to) the following anti obesity agents:
* Prescription drugs such as orlistat (Xenical), sibutramine (Meridia), and phentermine (Adipex-P, Celltech, Pro-Fast SA, Pro-Fast SR, Fastin, Oby trim, Zantryl, Teramine, Phentride, Phentercot, Obephen, Oby-cap); or
* Over-the-counter antiobesity agents (e.g., herbal supplements or other alternative remedies such as Cortislim, Dexatrim, Acutrim);
* Systemic steroids administered by oral, intravenous, or intramuscular route;
* Drugs that directly affect gastrointestinal motility (e.g., Reglan® and Propulsid®, and chronic [taken for more than 10 days within a 6-month period] macrolide antibiotics such as erythromycin and newer derivatives);
* Anti-depressants or benzodiazepines unless one of the following permitted drugs: escitalopram (Cipralex®), citalopram (Celexa®), clonazepam (Clonapam®), alprazolam (Xanax®), chlordiazepoxide (Librium®), diazepam (Valium®) and lorazepam (Ativan®);
* Calcitonin (e.g., Miacalcin®);
* Insulin;
* Exenatide (Byeta®);
* Sulfonylureas (e.g., Diamicron®, Amaryl®, Glucotrol®, Micronase®); or
* Meglitinides (e.g., Starlix®, Prandin®);
* Receipt of any investigational treatment (drug or device) within 90 days prior to screening; or
* Is an immediate family member of personnel directly affiliated with the study at the investigative sites, or is personally directly affiliated with the study at the investigative sites.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The change in body weight from Baseline to Week 16 | Week 16

SECONDARY OUTCOMES:
Rate of weight change | Week 16
Change in waist circumference from Baseline to Week 16 | Week 16
Changes from Baseline to Week 16 in measurements of obesity associated cardiovascular risk factors: sitting systolic and diastolic blood pressure, plasma lipid profile (LDL, non-HDL-C, TG, TC, and HDL-C), HbA1c, and FPG | Week 16
Change in the pharmacokinetic properties of olanzapine due to betahistine co-administration | Week 16
Change in psychiatric condition since randomization | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Yaffa Beck, Study Chair — OBEcure Ltd.
Locations (10):
- Canada (7):
  - Capital Health, Edmonton Mental Health Clinic, Edmonton, Alberta
  - Dr. Alexander McIntyre, Penticton, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Dr. Ivan Kowalchuk, Winnipeg, Manitoba
  - Capital District Health Authority, Halifax, Nova Scotia
  - Queen's University, Kingston, Ontario
  - Douglas Hospital Research Centre, Verdun (Montreal), Quebec
- Israel (3):
  - Abarbanel Hospital, Bat Yam
  - Geha Psychiatric Hospital, Petah Tikva
  - Lev Hasharon, Tirat Hacarmel